CLINICAL TRIAL: NCT05676918
Title: Maternal Well-being in the Postnatal Stage: Evaluation of Cognitive Biases and Validation of a Psychological Intervention
Brief Title: Maternal Well-being in the Postnatal Stage
Acronym: BIEMAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Universidad Pontificia de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCM-UPS-WELLBEING
Record Dates: First submitted 2022-11-10; First posted 2023-01-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Depression; Postpartum Disorder
MeSH Terms: conditions — Depression, Postpartum; Puerperal Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive Psychology Intervention (Experimental): Ten weekly sessions. Session duration: 90 minutes.
  Interventions: Behavioral: Positive Psychology Intervention
- Cognitive Behavior Therapy (Active Comparator): Ten weekly sessions. Session duration: 90 minutes.
  Interventions: Behavioral: Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — PPI includes 2 modules: hedonic well-being and eudaimonic well-being.
  Arms: Positive Psychology Intervention
Behavioral: Cognitive Behavior Therapy — CBT includes 3 modules: behavioral activation, cognitive restructuring, and interpersonal skills.
  Arms: Cognitive Behavior Therapy

SUMMARY:
The objective of this study is to design and validate an online intervention aimed at promoting well-being in women with postpartum depression. For this, the design of a multicomponent protocol consisting of empirically validated positive interventions and comparing these with a group Cognitive Behavioral Therapy (CBT) is proposed, following the National Institute for Health and Care Excellence (NICE) recommendations for the treatment of depression. Participants will be screened for inclusion in the program if they meet clinical criteria. After that, they will be randomly assigned to a CBT group or a positive psychology intervention (PPI) group.

DETAILED DESCRIPTION:
Participants will be randomly assigned to the CBT group or the PPI group. Both groups will be treated identically except for the type of intervention. Group assignment will be blind to both patients and investigators.

Both interventions have 10 weekly sessions. Sessions will be in groups and online.

CBT includes 3 modules: behavioral activation, cognitive restructuring, and interpersonal skills. Main contents (10 sessions): (1) Symptoms of Depression. Myths about motherhood. CBT approach; (2) Stress and Anxiety. Relaxation; (3 and 4) Increase pleasurable activities. Balance in life. To manage time; (5) Management of negative thoughts. Health concerns; (5 and 6) Increase positive thoughts; (7) social skills; (8) Communication skills and parner support; (9) Plan for the future. New routines and strategies; (10) Relapse prevention. CBT has been shown to be effective in reducing depressive symptoms and modifying attentional biases (Pearson et al., 2013).

On the other hand, a new protocol of positive interventions adapted for women after maternity (PPI) will be designed and applied. This multicomponent protocol includes interventions that have already been empirically validated in treating depression. PPI includes 2 modules: hedonic well-being and eudaimonic well-being. Main contents (10 sessions): (1) Symptoms of Depression. Myths about motherhood. PPI approach; (2) Mindfulness and positive emotions; (3) Gratitude and savoring; (4) Emotion regulation (5) Positive relationships and social support; (6) Compassion; (7) Personal strengths; (8) Goals and values; (9) Resilience; (10) Relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been mothers in the last year

Exclusion Criteria:

* Women who have been mothers in the last month,
* Women who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for substance abuse and/or dependence within 30 days prior to study participation,
* Women who have a serious mental disorder that makes it difficult to follow the protocol (e.g. serious neurocognitive problems or brain damage; schizophrenia and other psychotic disorders).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum depression change | Immediately before and after the intervention
  Edinburgh Postpartum depression scale (EPDS). Scores range from 0 to 30, where higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Positive and Negative Affect change | Immediately before and after the intervention
  Positive and Negative Affect Scale (PANAS). Positive emotions scores range from 10 to 50, where higher scores mean a better outcome. Negative emotions scores range from 10 to 50, where higher scores mean a worse outcome.
Satisfaction with life change (SWLS). Scores range from 5 to 35, where higher scores mean a better outcome. | Immediately before and after the intervention
  Satisfaction With Life Scale
Beliefs about pregnancy change | Immediately before and after the intervention
  The Pregnancy Related Beliefs Questionnaire (PRBQ-8). Scores range from 8 to 56. Higher scores indicate greater levels of dysfunctional attitudes towards motherhood.
Psychological well-being change | Immediately before and after the intervention
  Psychological well-being scale by Ryff (PWBS). PWBS-29 is composed for 29 items with a minumum score of 29 and a maximum score of 174. Self-acceptance scores range from 4 to 24; Positive Relationships with others scores range from 5 to 30; Autonomy scores range from 6 to 36; Environmental mastery scores range from 5 to 30; Purpose in life scores range from 5 to 30 and Personal Growth scores range from 4 to 24. Higher score in each subscale means a better outcome.
Maternal filial bond in the postpartum change | Immediately before and after the intervention
  The Postpartum Bonding Questionnaire (PBQ). Scores Range from 0 to 120. General factor scores range from 0 to 60 (Cut-off score 11= normal, 12 = high). Rejection of the infant scores range from 0 to 35. (cut-off 16 = normal, 17 = high). Infant-focused anxiety scores range from 0 to 10 (cut- off 9 = normal, 10 = high). Incipient abuse scores range from 0 to 10 ( cut-off 2 = normal, 3 = high). A high score in each factor indicates pathology.
Maternal self-efficacy change | Immediately before and after the intervention
  Maternal Self-efficacy Questionnaire (MSQ). Scores range from 10 to 40, where equal or greater scores than 31 means a high perception of maternal self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Covadonga Chaves, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Covadonga Chaves Vélez, Madrid, Pozuelo de Alarcón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Information on the evaluation and intervention protocol can be requested from the researchers. Likewise, the individual participant data can be provided on demand to guarantee the transparency of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Since the end of the study (June 2024) and for 10 years
Access Criteria: The individual participant data can be provided on demand to guarantee the transparency of the study.